CLINICAL TRIAL: NCT05961956
Title: A Proof-of-concept Study With NVDX3, an Osteogenic Implant of Human Allogenic Origin, in the Treatment of Low Grade Degenerative Lumbar Spondylolisthesis by Interbody Spine Fusion in Adults.
Brief Title: Study With NVDX3 for Treatment of Low Grade Degenerative Lumbar Spondylolisthesis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novadip Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVDX3-CLN02; 2022-002771-11 (EudraCT Number)
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Lumbar Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NVDX3 osteogenic implant (Experimental)
  Interventions: Drug: NVDX3

INTERVENTIONS:
Drug: NVDX3 — NVDX3 is implanted during a single surgical intervention.

SUMMARY:
Prospective, single arm, single-center clinical study to test NVDX3 in patients suffering from low grade one level degenerative lumbar (L1 - S1) spondylolisthesis. NVDX3 will be implanted during a single surgical intervention.

DETAILED DESCRIPTION:
This is a prospective, single arm, single-center PoC study in adult patients, suffering from a degenerative lumbar (L1-S1) spondylolisthesis, treated by spondylodesis in which NVDX3, an osteogenic implant from human allogeneic origin is used. The screening and implant surgery visits will be used as the reference timepoint respectively for the clinical and the radiological efficacy outcome evaluations.

As per standard of care, patients with DLS are followed up to 12 months post-intervention. In the context of this trial, patient safety and IMP efficacy will be followed up to 24 months post-implant surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years to ≤80 years.
2. Patient diagnosed with symptomatic DLS with confirmed:

   1. Classification: Meyerding grade I or II DLS
   2. One vertebral segment within the lumbar region from L1-S1
   3. Availability of AP and LAT X-ray, MRI and/or CT scan at which the diagnosis was made.
3. The estimated volume of targeted disc space to be filled (both inside and around the interbody cage) should not exceed 10cc.
4. Clinically meaningful pain or neurological symptoms with or without claudication confirmed by a preoperative ODI score >30, which have been unresponsive to a minimum of 3 consecutive months of structured conservative medical management (including at least pain medication, activity modification, and daily exercise).
5. Patient is eligible for surgery by minimally invasive or open transforaminal lumbar interbody fusion (TLIF)3.
6. Patient has understood and accepted to participate in the study according to all study procedures by signing the informed consent.

Exclusion Criteria:

1. History of previously attempted spinal fusion at the same vertebral level, or at a level immediately adjacent to the level intended to undergo the spondylodesis. Decompressive surgery alone (laminectomy) is not an exclusion criterion.
2. Patient with a BMI of ≥35.
3. Presence of clinically significant infection at the target implant site or presence of any systemic infection.
4. History of allergic reaction or any anticipated hypersensitivity to any of the following:

   1. Osteosynthesis materials (eg.cage, screws, rods,…),
   2. Anesthetic agents,
   3. Components of the NVDX3 implant
5. Presence of any auto-immune disease, with exception of well controlled diabetes type-1 or II, or auto-immune thyroid disorders.
6. Positive serology for human immunodeficiency virus (HIV), HBcAb and/or HBsAg.
7. Presence of an active tumor.
8. Documented metabolic bone disease or any disorder, such as but not limited to high-risk osteoporosis, that could interfere with the bone healing and bone metabolism.
9. Documented disease limiting mobility and functional assessments.
10. Chronic, ongoing, or planned use of medications that might affect bone metabolism or bone quality such as bisphosphonates, steroids, methotrexate, anticoagulants, immunosuppressants or immunotherapy.
11. Excessive smoking or history of chronic alcohol or drug abuse within the 12 months prior to screening
12. Use of any investigational drug within 60 days prior to screening.
13. Pregnant women or women of childbearing potential (WOCBP) not agreeing to use effective an effective method of birth control4 during the course of the study. Note: WOCBP including peri-menopausal women who have had a menstrual period within 1 year prior to surgery have to have a negative pregnancy test before entering in the study.
14. Any other psychosocial, mental and physical condition which, in the opinion of the investigator, could interfere with the trial conduct, the patient's compliance or influence interpretation of the results.
15. Patient with historically elevated radiation exposure levels that could in the opinion of the investigator introduce unacceptable radiation risks for the patient, when being accumulated with the radiological examinations planned in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Up to 24 months post implant surgery
  Description of all SAEs and NVDX3 related AEs

SECONDARY OUTCOMES:
Safety: all acute SAEs and NVDX3 related AEs | Between screening (V1) and 6 weeks post-IS (V4)
  Description of all acute SAEs and NVDX3 related AEs
Safety: all SAEs and NVDX3 related AEs | Beyond 6 weeks (V4 excluded) until 12 months post-IS
  Description of all SAEs and NVDX3 related AEs
Safety: all SAEs and NVDX3 related AEs | Beyond 12 months (V7 excluded) until 24 months post-IS
  Description of all SAEs and NVDX3 related AEs
Safety: TEAEs | a. Between screening and week 6 (V4 included) b. Between week 6 (V4 excluded) till month 12 (V7 included) c. Between month 12 (V7 excluded) till month 24 (V9 included) d. Full study duration
  Description of Treatment Emergent AEs (TEAEs)
Safety: related and unexpected (S)AEs | Between screening (v1) till 24 months post-IS
  Description of related and unexpected (S)AEs
Safety: AESI | Between screening (v1) till 24 months post-IS
  Description of AE of Special Interest (AESI)
Safety: Lab data | Between screening (v1) till 24 months post-IS
  Description of lab data
Safety: vital signs: physiological parameters | Between screening (v1) till 24 months post-IS
  Description of vital signs: body temperature, pulse rate, respiratory rate and blood pressure
Efficacy: Radiological assessments | a. 4 and 12 months post-IS based on CT compared to Hospital Discharge image acquisition and b. 24-months post-IS based on X-rays compared to the first post-operative X-ray acquisitions taken at 6 weeks post-IS
  Evaluate presence of cortical and trabecular bone formation
Efficacy: Radiological assessments | a. 4 and 12 months post-IS based on CT compared to Hospital Discharge image acquisition and b. 24-months post-IS based on X-rays compared to the first post-operative X-ray acquisitions taken at 6 weeks post-IS
  Evaluate presence of spinal fusion (Interbody/disc and facet joint fusion status)
Efficacy: Radiological assessments | At Hospital Discharge, 4 and 12 months post-IS
  Measure the average disc height variations based on CT
Efficacy: Clinical assessments: investigator questionnaire | At hospital discharge, 6 weeks, 4-, 6-, 12-, 18- and 24-months post-IS
  Physician rated Clinical Global Impression scale (CGI)
Efficacy: Clinical assessments: patient questionnaire | At hospital discharge, 6 weeks, 4-, 6-, 12-, 18- and 24-months post-IS
  Patient reported Functional assessments using the ODI
Efficacy: Clinical assessments: patient questionnaire | At hospital discharge, 6 weeks, 4-, 6-, 12-, 18- and 24-months post-IS
  Patient reported Numeric rating scale (NRS) for pain

CONTACTS AND LOCATIONS:
Overall Officials: David BREUSKIN, MD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (1):
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg